CLINICAL TRIAL: NCT00961636
Title: A Worldwide, Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Evaluate the Long-term Efficacy, Safety and Tolerability of ERN/LRPT in Patients With Dyslipidemia
Brief Title: A Long-term Study of ERN/LRPT (Extended Release Niacin/Laropiprant [MK0524A]) in Patients With Dyslipidemia (0524A-102)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-102; 2009_634
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ERN/LRPT (Experimental): One 1g/20 mg tablet ERN/LRPT once daily for 4 weeks, then two 1g/20 mg
  tablets daily (2g/40 mg total) for 28 weeks
  Interventions: Drug: ER niacin (+) laropiprant (ERN/LRPT)
- ERN/LRPT then ERN (Experimental): One 1g/20mg tablet ERN/LRPT once daily for 4 weeks, then two 1g/20 mg tablets daily (2g/40 mg total) for 16 weeks then Two 1g tablets ERN (2g total) once daily for 12 weeks.
  Interventions: Drug: ER niacin (+) laropiprant (ERN/LRPT); Drug: Extended-release niacin (ERN)
- Placebo (Placebo Comparator): One tablet placebo to ERN/LRPT once daily for 4 weeks, then two tablets placebo to ERN/LRPT daily for 28 weeks.
  Interventions: Drug: Placebo to ERN/LRPT

INTERVENTIONS:
Drug: ER niacin (+) laropiprant (ERN/LRPT) — One 1g/20 mg tablet ERN/LRPT once daily for 4 weeks, then two 1g/20 mg tablets daily (2g/40 mg total) for 28 weeks
  Arms: ERN/LRPT
Drug: ER niacin (+) laropiprant (ERN/LRPT) — One 1g/20mg tablet ERN/LRPT once daily for 4 weeks, then two 1g/20 mg tablets daily (2g/40 mg total) for 16 weeks.
  Arms: ERN/LRPT then ERN
Drug: Extended-release niacin (ERN) — Two 1g tablets ERN (2g total) once daily for 12 weeks.
  Arms: ERN/LRPT then ERN
Drug: Placebo to ERN/LRPT — One tablet placebo to ERN/LRPT once daily for 4 weeks, then two tablets placebo to ERN/LRPT daily for 28 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of laropiprant (LRPT) to reduce flushing symptoms beyond 6 months and will measure the impact of withdrawal of laropiprant in patients following 20 weeks of stable maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male, or a female who is unlikely to conceive, as indicated by meeting at least one of the following conditions: (a) Patient is a male.(b) Patient is a female of reproductive potential and either agrees to remain abstinent (if this form of birth control is accepted by local regulatory agencies and review committees as the sole method of birth control) or use (or have their partner use) 2 acceptable methods of birth control within the projected duration of the study.(c) Patient is a female who is not of reproductive potential and therefore eligible to participate in this study without requiring the use of contraception.
* Lipid-modifying therapy (LMT) is appropriate for the patient
* Patient meets one of the following criteria based on the National Cholesterol Education Program Adult Treatment Panel III guidelines : 1) High risk and is on a statin with LDL-cholesterol (LDL-C) <100 mg/dL or intolerant to statins with LDL-C <120 mg/dL; 2) Multiple risk with LDL-C <130 mg/dL; 3) Low risk with LDL-C <190 mg/dL
* Patient has triglyceride levels <500 mg/dL

Exclusion Criteria:

* Patient is pregnant, breast-feeding, or expecting to conceive
* Patient has a history of cancer within 5 years of screening (except certain skin and cervical cancers)
* Female patient plans to donate eggs during the study
* Male patient plans to donate sperm during the study
* Patient has or has a history of any condition, therapy, or lab abnormality that might confound the study results, interfere with participation for the full duration of the study, or make participation in the study not in the patient's best interest
* Patient has donated or received blood within 8 weeks of screening or plans to donate/receive blood during and 8 weeks after the study
* Patient is experiencing menopausal hot flashes
* Patient has chronic heart failure, uncontrolled cardiac arrhythmias, or poorly controlled hypertension
* Patient has type 1 or 2 diabetes and is poorly-controlled, newly diagnosed, has recently had repeated hypoglycemia, or is taking new or recently adjusted antidiabetic medication
* Patient has uncontrolled metabolic or endocrine disease that influences serum lipids or lipoproteins
* Patient has kidney disease
* Patient had active peptic ulcers within 3 months of screening
* Patient has a history of heart attack, stroke, heart bypass surgery, angina, or angioplasty within 3 months of screening
* Patient is human immunodeficiency virus (HIV) positive
* Patient is taking or has taken niacin >50 mg daily within 6 weeks of screening
* Patient has had a change to type or dose of LMT regimen within 6 weeks of Visit 1
* Patient is taking a statin and a fibrate at screening
* Patient is taking a long acting non-steroidal anti-inflammatory drug (NSAID), such as naproxen or aspirin >100 mg per day at screening
* Patient has arterial bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Maccubbin DL, Chen F, Anderson JW, Sirah W, McCrary Sisk C, Kher U, Olsson AG, Bays HE, Mitchel YB. Effectiveness and safety of laropiprant on niacin-induced flushing. Am J Cardiol. 2012 Sep 15;110(6):817-22. doi: 10.1016/j.amjcard.2012.05.009. Epub 2012 Jun 8. PMID 22683042

RESULTS

PARTICIPANT FLOW:
Groups:
- ERN/LRPT: One 1g/20 mg tablet Extended -release niacin (+) laropiprant (ERN/LRPT) once daily for 4 weeks, then two 1g/20 mg tablets daily (2g/40 mg total) for 28 weeks
Period: Overall Study
Arm/Group | ERN/LRPT | ERN/LRPT Then ERN | Placebo
Started | 463 | 456 | 233
Completed | 356 | 325 | 201
Not Completed | 107 | 131 | 32
Not completed — Adverse Event | 35 | 54 | 13
Not completed — Flushing Symptoms | 29 | 46 | 3
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Physician Decision | 3 | 1 | 1
Not completed — Protocol Violation | 9 | 5 | 1
Not completed — Withdrawal by Subject | 29 | 22 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERN/LRPT | ERN/LRPT Then ERN | Placebo | Total
Number analyzed (Participants) | 463 | 456 | 233 | 1152
Age, Customized [Number; unit: Participants]
  < 65 years | 334 | 328 | 166 | 828
  >=65 years | 129 | 128 | 67 | 324
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 144 | 87 | 415
  Male | 279 | 312 | 146 | 737

OUTCOME MEASURES:

1. Primary Outcome: Number Participants With Days Per Week With Global Flushing Severity Score (GFSS) ≥4 Partitioned Into 6 Categories During the Postwithdrawal Period
Description: Flushing symptoms were recorded using participant's response to the Global Flushing Severity Score (GFSS), which assessed the overall severity of the flushing experience, using a scale of 0 (no symptom) to 10 (extreme). The number of days/week was derived as: 7*(total number of days with GFSS ≥4 across Weeks 21-32 divided by the total number of days with nonmissing GFSS across the same period). The number of days/week with a GFSS ≥4 for each participant was listed in 1 of the following 6 categories: 0, >0 to 0.5, >0.5 to 1, >1 to 2, >2 to 3, and >3 days per week.
Time Frame: Week 21 to Week 32
Population: Analysis performed using the Full Analysis Set (FAS) population which included all randomized participants that did not have a withdrawal visit and/or did not have at least 1 GFSS score during the post-withdrawal period (Weeks 21 to 32).
Measure: Number; unit: Participants
Arm/Group | ERN/LRPT | ERN/LRPT Then ERN | Placebo
Number analyzed (Participants) | 362 | 354 | 207
Participants
  0 Days per week | 291 | 181 | 188
  >0 to ≤ 0.5 Days per week | 43 | 74 | 7
  >0.5 to ≤1 Days per week | 3 | 32 | 4
  >1.0 to ≤2 Days per week | 8 | 30 | 3
  >2 to ≤3 Days per week | 1 | 17 | 1
  >3 Days per week | 16 | 20 | 4
Statistical Analysis 1: Comparison: ERN/LRPT vs ERN/LRPT Then ERN; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The closed ordered testing procedure was applied to the efficacy hypotheses. If statistical significance was achieved for the primary hypothesis, then the secondary hypothesis was tested. All tests were performed at significance level 0.05; Cochran-Mantel-Haenszel (CMH) test was stratified by country

2. Secondary Outcome: Number of Participants With Maximum GFSS ≥4 During the Post-withdrawal Period
Description: Flushing symptoms were recorded using participant's response to the Global Flushing Severity Score (GFSS), which assesses the overall severity of the flushing experience (including redness, warmth, tingling, or itching) using a scale with response categories of None, Mild, Moderate, Severe, and Extreme. The categories were supplemented with numbers 0 to 10 to allow for greater precision within each category (None=0, Mild=1-3, Moderate=4-6, Severe=7-9, Extreme=10). The daily response was recorded in the morning, and reflected the symptoms experienced during the previous 24 hours.
Time Frame: Week 21 to Week 32
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ERN/LRPT | ERN/LRPT Then ERN | Placebo
Number analyzed (Participants) | 362 | 354 | 207
Participants | 71 | 173 | 19
Statistical Analysis 1: Comparison: ERN/LRPT vs ERN/LRPT Then ERN; Test type: Superiority or Other; p < 0.001, Unconditional Miettinen and Nurminen — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Of 1152 randomized participants, 1148 participants took at least one dose of study medication and were included in the analyses of safety.
Arm/Group | ERN/LRPT | ERN/LRPT Then ERN | Placebo
Serious Adverse Events (participants affected / at risk) | 17/461 | 34/455 | 13/232
Other Adverse Events (participants affected / at risk) | 136/461 | 162/455 | 37/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERN/LRPT (N=461) | ERN/LRPT Then ERN (N=455) | Placebo (N=232)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epileptic aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERN/LRPT (N=461) | ERN/LRPT Then ERN (N=455) | Placebo (N=232)
Nasopharyngitis (Infections and infestations) | 33 (40) | 34 (35) | 11 (12)
Paraesthesia (Nervous system disorders) | 23 (53) | 28 (65) | 6 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 51 (67) | 66 (116) | 17 (18)
Flushing (Vascular disorders) | 52 (77) | 85 (130) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications derived from this study should include input from the investigator(s) and Sponsor personnel. Subsequent to the multicenter publication, or 24 months after completion of the study, whichever comes first, an investigator and/or his/her colleagues may publish the results for their study site independently. The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.